CLINICAL TRIAL: NCT01819285
Title: Phase III Comparison of Early vs Delayed Endocrine Manipulation (Orchiectomy or LHRH Agonist Therapy) in Previously Untreated Patients With Nonmetastatic Asymptomatic Carcinoma of the Prostate
Brief Title: Early Compared With Delayed Hormone Therapy in Treating Patients With Nonmetastatic Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-30891
Record Dates: First submitted 2013-03-18; First posted 2013-03-27 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Neoplasm, Prostate
Keywords: Malignant Neoplasm of Prostate; Tumor-node-metastasis (TNM) Staging Regional Lymph Nodes (N0-2); Not suitable for local treatment with curative intent
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (2):
- Immediate Endocrine Therapy (Active Comparator): Immediate Endocrine Therapy. Orchiectomy or LHRH Agonist Therapy plus (initially) Antiandrogen Therapy. Buserelin (BSRL); Cyproterone acetate (Androcur) (CPTR), Cyproterone acetate (Androcur)(NSC-81430). Treatment initiated within 1 month of randomization.
  Interventions: Procedure: Immediate Orchiectomy or depot LHRH
- Delayed Endocrine Therapy (Experimental): Orchiectomy or LHRH Therapy plus (initially) Antiandrogen Therapy. BSRL; CPTR. Treatment delayed until onset of symptoms.
  Interventions: Procedure: Delayed Orchiectomy or depot LHRH

INTERVENTIONS:
Procedure: Immediate Orchiectomy or depot LHRH
  Arms: Immediate Endocrine Therapy
Procedure: Delayed Orchiectomy or depot LHRH
  Arms: Delayed Endocrine Therapy

SUMMARY:
Objectives

I. Compare, in a randomized Phase III multi-institutional setting, symptom-free survival time of patients with asymptomatic carcinoma of the prostate (T0-4, N0-2, M0) not suited for local curative treatment who are randomly assigned to immediate vs. delayed endocrine intervention (orchiectomy or luteinizing hormone releasing hormone (LHRH) agonist therapy).

II. Compare the overall survival of these two groups of patients.

III. Compare the time to first evidence of distant progression (N4 or M1) of these two treatment groups.

IV. Evaluate the prognostic significance of pretreatment laboratory data and monitor these parameters following endocrine therapy.

V. Study the prognosis of various sub-groups of patients stratified according to performance status, local tumor extent, nodal status, and choice of endocrine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven, newly diagnosed asymptomatic (with the exception of voiding disturbances) carcinoma of the prostate T0-4 N0-2 M0 which is not suitable for local treatment with curative intent (radical prostatectomy, radiation therapy).
* All T stages are acceptable (UICC 1982). The stage is determined by rectal palpation.
* Patients with regional lymph node metastases smaller than 5 cm (N0-2), determined either by CT or ultrasonography, preferable with cytologic confirmation.
* Life expectancy of at least six months.
* WHO performance status score 0-1.
* Informed consent. Patients must be prepared to undergo an orchiectomy or continuous treatment with a depot LHRH analogue.
* Continuous follow-up until death if possible.

Exclusion Criteria:

* Other malignancies diagnosed during the last 10 years, apart from treated basal cell carcinoma of the skin.
* Prostate cancer known for longer than one month before entering the study.
* Pain caused by the prostate cancer or its metastases.
* Any previous treatment for prostate cancer (radical prostatectomy, radiation therapy, endocrine treatment, etc.) Note: TUR-P for voiding disturbances is allowed at any time and is not an exclusion criterion.
* Patients with ureteric obstruction caused by local infiltration of prostatic cancer and other evidence of locally advanced disease which could cause fatal complications if untreated (e.g. rectal stenosis, thrombosis of pelvic veins).
* Patients with palpable or juxtaregional lymph node metastasis (paraaortic, supraclavicular, inguinal, N3-4).
* Patients with evidence of distant metastases (bone, lung, liver).
* Age over 80 years. Performance status WHO score 2, 3 and 4 (any reason).
* Patient who refuses orchiectomy or longterm subcutaneous implants of LHRH analogue in two monthly intervals.

Expected difficulties with follow-up for any reason.

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 985 (Actual)
Dates: Start 1990-02; Primary Completion 2004-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | 13 years from first patient in

SECONDARY OUTCOMES:
Overall symptom free survival time | 13 years from first patient in
Time until first evidence of distant progression | 13 years from first patient in
Prognostic importance of pretreatment laboratory data | 13 years from first patient in
  prostate cancer mortality and overall mortality according to pretreatment laboratory data
Prognosis of particular sub-groups | 13 years from first patient in
  prostate cancer mortality and overall mortality according to particular sub-groups (following stratification factors): performance status (0 vs 1), the local tumor extent (T0-2 vs T3-4), nodal status (N0 vs N1-2), the choice of hormonal therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Urs Studer, MD, Study Chair — Insel Gruppe AG, University Hospital Bern

REFERENCES:
- [Derived] Studer UE, Whelan P, Wimpissinger F, Casselman J, de Reijke TM, Knonagel H, Loidl W, Isorna S, Sundaram SK, Collette L; EORTC Genitourinary Cancer Group. Differences in time to disease progression do not predict for cancer-specific survival in patients receiving immediate or deferred androgen-deprivation therapy for prostate cancer: final results of EORTC randomized trial 30891 with 12 years of follow-up. Eur Urol. 2014 Nov;66(5):829-38. doi: 10.1016/j.eururo.2013.07.024. Epub 2013 Jul 24. PMID 23932338
- See also: Related Info — http://www.eortc.be/clinicaltrials/details.asp?protocol=30891